CLINICAL TRIAL: NCT02812069
Title: WarmSmart Warming Protocol
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety issue
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-942
Record Dates: First submitted 2016-05-19; First posted 2016-06-23 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- minor to moderate surgical procedure (Other): The ThermaZone® Device will be used for 30 minutes to warm the cervical spine during
  Interventions: Device: ThermaZone® Device

INTERVENTIONS:
Device: ThermaZone® Device — The device will be used to intraoperatively warm patients having minor-to moderate surgical procedures

SUMMARY:
Hypothermia during surgery and in the postoperative period is associated with adverse outcomes including impaired drug metabolism, cardiac morbidity, shivering, impaired immune function, coagulopathy, and increased use of hospital resources. Several clinical studies have demonstrated that maintenance of normothermia during the perioperative period significantly reduces morbidity.

Mercury Biomed has developed a patient-warming system, WarmSmart, that potentially transfers adequate heat through hands and feet based on the physiological principle of peripheral arterio-venous shunt vaso-dilation. The technology works as a two-step process by selective thermal stimulation along the spinal cord to up-regulate blood flow to arterio-venous shunts and triggering arterio-venous shunt vasodilation and by applying circulating water heat exchangers to the palmar and plantar glabrous skin to warm highly perfused shunts in that area.

General anesthesia reduces the vasoconstriction threshold (triggering core temperature) by 1-2°C, thus promoting arteriovenous shunt dilation. It remains unknown, though, whether cervical spine warming further augments arterio-venous shunt dilation during general anesthesia. If spine heating proves unnecessary under anesthesia, Mercury Biomed's WarmSmart warming could be simpler and less expensive. Investigators therefore propose to test the hypothesis that cutaneous heating near the cervical spine does not further augment arterio-venous flow in fingers during general anesthesia.

Investigators propose to enroll ten patients. The patients will be pre-warmed and warmed intraoperatively with forced-air to maintain a core temperature near 36°C.

A ThermaZone® Device capable of heating the cervical spine area will be positioned behind the patient's neck upon arrival in the operating rooms. Additionally a forced-air warmer will be positioned appropriately and activated as soon as practical, usually after prepping and draping. Ambient temperature will be maintained near 20°C.

After about one hour of anesthesia when temperature and other factors are stable, investigators will start a 30-minute observation period. Thereafter investigators will activate the cervical spine warming system for 30 minutes (warming measurement period) and thereafter have a 30 minutes control period again.

Measurements will be recorded such as mean-skin temperature, distal esophageal temperature, MAC fraction, mean-arterial pressure and finger blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. Body-mass index 20-33 kg/m2;
2. Age 18-70 yrs;
3. ASA Physical Status 1-3.

Exclusion Criteria:

1. Serious skin lesions on the hands or arms;
2. History of serious vascular disease in the arms, including Raynaud's Syndrome;
3. Pre-operative fever or infection;
4. Surgery expected to be supine and in neutral position.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
volume plethysmography | Recorded from the time the ThermaZone® Device is placed for 30 minutes to thirty minutes after it's removal at 10-minute intervals from the beginning of the initial observation period until the end of the post-warming recovery period.
mean-skin temperature | Recorded from the time the ThermaZone® Device is placed for 30 minutes to thirty minutes after it's removal at 10-minute intervals from the beginning of the initial observation period until the end of the post-warming recovery period.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, M.D., Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No